CLINICAL TRIAL: NCT05788120
Title: Incidence and Morbidity of Cardiac Rhythm Disorders in Patients Assisted by Extra Corporeal Membrane Oxygenation Veno-arterial (ECMO VA) for Refractory Cardiogenic Shock
Brief Title: Incidence and Morbidity of Cardiac Rhythm Disorders in Patients Assisted by ECMO-VA for Refractory Cardiogenic Shock
Acronym: CAVA-ECMO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221056
Record Dates: First submitted 2023-03-06; First posted 2023-03-28 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Rhythm Disorder
Keywords: Arrhythmia; Veno-arterial Extra Corporeal Membrane; Oxygenation (VA ECMO); Cardiogenic shock.
MeSH Terms: conditions — Arrhythmias, Cardiac; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with refractory cardiogenic shock assisted with ECMO VA
  Interventions: Other: Follow up by phone call

INTERVENTIONS:
Other: Follow up by phone call — Centralized review of ECGs by the Pitié-Salpêtrière rhythmology department and collection of vital status at 12 months (if information not available, telephone call to the patient)

SUMMARY:
Brief Summary : Rhythm disorders are a frequent and potentially serious complication of critical patients in the ICU and postoperative cardiac surgery. In particular, atrial fibrillation (AF) is the most common rhythm disorder in patients admitted to the ICU and is associated with excess mortality during acute circulatory failure. In postoperative cardiac surgery, AF affects 15 to 45% of patients. In addition to hemodynamic effects, AF increases the risk of stroke, bleeding, respiratory or renal failure, and doubles mortality at 30 days and 6 months. In the longer term, the recurrence rate of AF within 1 year after hospital discharge is about 50%. Similarly, other rhythm disorders, supraventricular or ventricular, can be life-threatening in ICU patients.

While the incidence and complications of rhythm disorders are well documented during sepsis, cardiogenic shock or after cardiac surgery, there are to our knowledge no data on the frequency and complications of rhythm disorders in patients assisted by VA ECMO.

The primary objective is to describe the incidence of supraventricular rhythm disorders in patients assisted by VA ECMO.

DETAILED DESCRIPTION:
This study is an observational study to describe the conditions of occurrence of arrhythmias, particularly atrial fibrillation, in patients supported by VA ECMO, as well as their short-term and long-term prognosis. Patients will be recruited from the intensive care units and CRFs will be completed by the investigators at each of the participating centers. Data will be collected directly from the medical records, except for vital status at 1 year, which may be collected by telephone from the patient by the investigator at the center in the absence of data in the medical record.

Atrial fibrillation episodes will be recorded on a 12-lead electrocardiogram and securely transmitted to the coordinating center. In addition, investigators will send weekly data to the principal investigator for incidence calculation. Patients or their relatives will be informed about the study by an information sheet presented and explained by the investigator or another person authorized to conduct the research. The investigator will record the patient's consent in the patient's medical record.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Assistance with VA ECMO

Exclusion Criteria:

* Opposition to the use of data.
* Persons under legal protection (curators, guardianship), judicially safeguarded.
* VA ECMO for refractory cardiac arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major Patients Assisted by VA ECMO in Intensive care
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2027-04-28 (Estimated); Study Completion 2027-04-28 (Estimated)

PRIMARY OUTCOMES:
Number of atrial fibrillation in patients assisted by veno-arterial ECMO. | day 30
  Atrial fibrillation will be defined as an episode of AF ≥ 30 minutes or requiring pharmacological or electrical cardioversion.

SECONDARY OUTCOMES:
Number of ventricular rhythm disorders | day 30
  ventricular tachycardia, ventricular fibrillation
duration of VA ECMO support | day 30
  duration of VA ECMO support
duration of ICU stay | day 30
  duration of ICU stay
duration of mechanical ventilation | day 30
  duration of mechanical ventilation
Number of living patient | day 28, day 360
  Number of living patient
Number of thrombo-embolic complications | day 30
  acute limb ischemia, circuit thrombosis, membrane thrombosis
Number of neurological complications | day 30
  ischemic and hemorrhagic stroke
Number of bleeding complications | day 30
  bleeding requiring transfusion of packed red blood cells (> 3 units / 24h) or requiring surgical intervention or interventional procedure (digestive or implantation site bleeding, need for revision surgery

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Angers, Angers
  - Hospices Civils de Lyon - Hôpital Louis Pradel, Bron
  - CHU Caen Normandie - Hôpital Côte de Nacre, Caen
  - CHRU Tours - Hôpital Trousseau, Chambray-lès-Tours
  - CHU Dijon Bourgogne - Hôpital François Mitterrand, Dijon
  - CHU Grenoble Alpes - Site Nord, Grenoble
  - CHU Lille - Institut Cœur Poumon, Lille
  - CHU Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU Nantes - Hôpital Nord Laennec, Nantes
  - Pitié Salpêtrière Hospital, Intensive Care Unit - Resuscitation, Paris
  - Pitié-Salpêtrière Hospital, Cardiovascular Surgery Intensive Care Unit, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Bichat, Paris
  - CHU Bordeaux - Hôpital cardiologique, GH Sud Pessac, Pessac
  - CHU Rennes, Hôpital Pontchaillou, Rennes
  - Hôpitaux universitaires de Strasbourg - Hôpital Civil, Strasbourg
  - CHU Toulouse - Hôpital de Rangueil, Toulouse
  - CHRU Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal